CLINICAL TRIAL: NCT00975962
Title: New Acute Treatment for Stroke - The Effect of Remote PERconditioning
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: TRYG Foundation (Other); Aase and Ejnar Danielsens Foundation (Other); Danish National Research Foundation (Other)
Responsible Party: Grethe Andersen M.D doctor, Department of Neurology Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VEK 19752
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Acute Stroke
Keywords: Stroke; Neuroprotection; remote preconditioning; Salvage index (%): Difference in infarct growth (PWI-DWI)
MeSH Terms: conditions — Stroke | interventions — Tissue Plasminogen Activator; Fibrinolytic Agents

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thrombolysis + Remote perconditioning (Experimental): Remote perconditioning (rIPerC) undertaken in ambulance on rute to hospital in case of suspected stroke.
  The rIPerC consists of 4 cycles of 5 minute total occlusion of blood flow to the non-paretic arm separated by 5 minutes of reperfusion. The occlusion is secured by inflating a standard blood pressure cuff to 25 mmHg above the systolic blood pressure. Written instruction on cuff inflation and paramedic's documentation of their procedure were written in a standard report which was turned over to a study nurse upon arrival to the hospital, and filed. The investigators were hence blinded to the prehospital rIPerC.
  Interventions: Procedure: Thrombolysis + remote perconditioning
- Thrombolysis (Active Comparator): Thrombolysis without pretreatment with remote perconditioning
  Interventions: Drug: Actilyse

INTERVENTIONS:
Drug: Actilyse — Actilyse according to guidelines without pretreatment with remote persconditioning
  Arms: Thrombolysis
Procedure: Thrombolysis + remote perconditioning — The rIPerC consists of 4 cycles of 5 minute total occlusion of blood flow to the non-paretic arm separated by 5 minutes of reperfusion. The occlusion is secured by inflating a standard blood pressure cuff to 25 mmHg above the systolic blood pressure. Written instruction on cuff inflation and paramedic's documentation of their procedure were written in a standard report which was turned over to a study nurse upon arrival to the hospital, and filed. The investigators were hence blinded to the prehospital rIPerC.
  Arms: Thrombolysis + Remote perconditioning

SUMMARY:
This study is a blinded randomized study. Randomization for treatment/not treatment with remote perconditioning takes place during transportation to the hospital. This is because the investigators' hypothesis states that remote perconditioning is neuro-protective and the effect is proportionally larger with early treatment. As the size of the effect is unknown, the investigators will use multiple magnetic resonance imaging (MRI) scans to determine the size of a potential neuro-protective effect.

The aims of this study are:

1. To describe method of remote perconditioning in clinical practice regarding feasibility. Pros and cons and potential limitations.
2. To estimate the size of the effect of remote perconditioning in combination with recombinant tissue plasminogen activator (rtPa) treatment within four and a half hours of onset of symptoms.

DETAILED DESCRIPTION:
Final inclusion and informed consent takes place after first MRI in patients eligible for rtPA.

Follow-up MRI after 24h and 1 month. Clinical outcome at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Significant ischemic stroke suspicion (NIHSS 1-24) and paresis of an extremity.
* Treatment with rtPa within 4.5 hours from debut of symptoms.
* Age above 18 (changed from 01.01.2010 to no upper age limit)
* Independent in daily living before the acute onset of symptoms. (mrs</=2)
* MR scan showing DWI lesion, consistent with acute ischemic stroke.

Exclusion Criteria:

* Contraindications for iv rtPA
* Onset of symptoms older than 4.5 hours
* Previous diseases of the brain: Intracranial aneurisms or arteriovenous malformations. Brain surgery or hemorrhagic stroke. Former ischemic stroke within the last 3 months.
* Heart diseases: Infectious endocarditis or suspicion of septic emboli, pericarditis, ventricular thrombosis, aneurisms of the heart wall or major heart failure.
* Serious diseases: Cancer, AIDS, dementia, significant abuse, renal failure, liver diseases such as liver failure, cirrhosis, portal hypertension, active hepatitis.
* Pregnancy
* Major ischemic stroke where the patient is unconscious.(NIHSS > 25).
* Symptoms suspect for migraine, Multiple sclerosis, TIA or another neurological disease than ischemic stroke.

MR scan:

* Contraindications for MRI scans
* Tumor cerebri, cerebral abscesses
* Known hypersensitivity to Gadovist or any of its ingredients, acute or chronic severe renal impairment (GFR < 30 ml/min/1.73m2), acute renal insufficiency of any severity due to the hepato-renal syndrome or in the perioperative liver transplantation period.
* Caution with using Gadovist to patients with severe cardiovascular disease, and only to be used after a risk-benefit assessment.
* Caution with using Gadovist in patients with low threshold for seizures.

Lab data:

* Blood glucose < 2, 8 mmol/l or > 22 mmol/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Salvage index (%): Difference in infarct growth (PWI-DWI) after 24 hours among patients treated with preconditioning and those not treated. | February 2012

SECONDARY OUTCOMES:
Final size of the infarct (T2 MRI after 1 month). Final infarct size adjusted after prognostic factors. | February 2012

CONTACTS AND LOCATIONS:
Overall Officials: Grethe Andersen, M.D Doctor, Principal Investigator — Department of Neurology Aarhus University Hospital
Locations (1):
- Department of Neurology, Aarhus University Hospital, Aarhus, Aarhus, Denmark

REFERENCES:
- [Derived] Hougaard KD, Hjort N, Zeidler D, Sorensen L, Norgaard A, Hansen TM, von Weitzel-Mudersbach P, Simonsen CZ, Damgaard D, Gottrup H, Svendsen K, Rasmussen PV, Ribe LR, Mikkelsen IK, Nagenthiraja K, Cho TH, Redington AN, Botker HE, Ostergaard L, Mouridsen K, Andersen G. Remote ischemic perconditioning as an adjunct therapy to thrombolysis in patients with acute ischemic stroke: a randomized trial. Stroke. 2014 Jan;45(1):159-67. doi: 10.1161/STROKEAHA.113.001346. Epub 2013 Nov 7. PMID 24203849